CLINICAL TRIAL: NCT01090895
Title: Effect of Vitamin C Infusion on Coronary Reperfusion Indexes
Brief Title: Treatment of Reperfusion Event by Vitamin C Infusion
Acronym: TREVI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Full professor of internal medicine, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Violi012009
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Angina Pectoris
Keywords: Percutaneous Coronary Intervention; Vitamin C; Biomarkers; Magnetic Risonance
MeSH Terms: conditions — Angina Pectoris | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin C (Active Comparator): Vitamin C infusion
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — Intravenous infusion of vitamin C (1 g) 10 minutes before percutaneous coronary intervention.
  Other Names: Ascorbic Acid
  Arms: Vitamin C
Drug: Placebo — Intravenous infusion of placebo(saline solution) 10 minutes before percutaneous coronary intervention.
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
Primary Hypothesis: Prophylactic Vitamin C Intravenous Infusion at the time of percutaneous coronary intervention (PCI) would limit the size of the infarct, assessed by measurements of cardiac biomarkers, during acute myocardial infarction.

Secondary Hypotheses: Prophylactic Vitamin C Intravenous Infusion at the time of percutaneous coronary intervention (PCI) would limit the size of the infarct, as measured by the area of delayed hyperenhancement that was seen on cardiac magnetic resonance imaging (MRI), assessed on day 5 after infarction, during acute myocardial infarction.

DETAILED DESCRIPTION:
This is a multicenter, prospective, controlled, randomized study that will be conducted at up to 5 centers in Italy. All patients who meet the eligibility criteria will be randomized to receive during surgical procedure an intravenous infusion of Vitamin C or Placebo.

Patients will have repeat clinical follow-up to 5 days, 3 and 6 months and 1 year.

The new angiography evaluation will be done if necessary. The study population will consist of at least 100 patients who presented within 12 hours after the onset of chest pain, who had ST-segment elevation of more than 0.1 mV in two contiguous leads, and for whom the clinical decision was made to treat with percutaneous coronary intervention (PCI). Following confirmation of eligibility criteria, patients will be randomized in a 1:1 ratio to receive prophylactic infusion of Vitamin C or Placebo. The coronary angiograms will be assessed at a core laboratory with Quantitative Coronary Angiography.

The incidence of clinical events, including death, myocardial infarction, target vessel revascularization, stent thrombosis, will be evaluated at 1, 3, 6 and, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who presented within 12 hours after the onset of chest pain, who had ST-segment elevation of more than 0.1 mV in two contiguous leads, and for whom the clinical decision was made to treat with percutaneous coronary intervention (PCI)
* Patients will be eligible for the study whether they were undergoing primary PCI.
* Signed written informed consent

Exclusion Criteria:

* Patients with cardiac arrest, ventricular fibrillation, cardiogenic shock, stent thrombosis, previous acute myocardial infarction, or angina within 48 hours before infarction were not included in the study
* Patients with evidence of coronary collaterals (2-3 Rentrop) to the region at risk on initial coronary angiography (at the time of admission) will be excluded
* The patient has impaired renal function (creatinine > 3.0 mg/dl)
* The patient has known allergies to aspirin, clopidogrel bisulfate and ticlopidine, heparin, contrast media or stainless steel that cannot be managed medically
* The patient needs therapy with warfarin
* The patient has a life expectancy less than 12 months
* Recipient of heart transplant
* The patient is currently participating in an investigational drug or another device study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Specific key observations used to measure the effect of experimental treatment in this study are the incidence of Major Adverse Cardiovascular Events. | 12 months
  Cardiovascular Death, Myocardial Infarction, Stent Thrombosis, Repeat Revascularization, Stroke, Transient Ischemic Attack

SECONDARY OUTCOMES:
Myocardial damage and microcoronary disfunction by cardiac magnetic resonance imaging | 7 days
  Prophylactic Vitamin C Intravenous Infusion at the time of percutaneous coronary intervention (PCI) would limit the size of damage within 7 days after PCI.
Improvement of reperfusion indexes (corrected Thrombolysis In Myocardial Infarction frame count and myocardial blush grade) | post PCI
  Prophylactic Vitamin C Intravenous Infusion at the time of percutaneous coronary intervention (PCI) could improve the reperfusion indexes.
Early incidence of Major Adverse Cardiovascular Events. | 1 month
  Cardiovascular Death, Myocardial Infarction, Stent Thrombosis, Repeat Revascularization, Stroke, Transient Ischemic Attack
Late incidence of Major Adverse Cardiovascular Events. | 3 months
  Cardiovascular Death, Myocardial Infarction, Stent Thrombosis, Repeat Revascularization, Stroke, Transient Ischemic Attack

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, Full Prof, Study Chair — Divisione di Prima Clinica Medica - Sapienza University of Rome
Locations (1):
- Sapienza Università di Roma, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pignatelli P, Sanguigni V, Paola SG, Lo Coco E, Lenti L, Violi F. Vitamin C inhibits platelet expression of CD40 ligand. Free Radic Biol Med. 2005 Jun 15;38(12):1662-6. doi: 10.1016/j.freeradbiomed.2005.02.032. Epub 2005 Mar 23. PMID 15917194
- [Background] Cordova C, Musca A, Violi F, Perrone A, Alessandri C. Influence of ascorbic acid on platelet aggregation in vitro and in vivo. Atherosclerosis. 1982 Jan;41(1):15-9. doi: 10.1016/0021-9150(82)90064-8. PMID 7073791
- [Background] Basili S, Tanzilli G, Mangieri E, Raparelli V, Di Santo S, Pignatelli P, Violi F. Intravenous ascorbic acid infusion improves myocardial perfusion grade during elective percutaneous coronary intervention: relationship with oxidative stress markers. JACC Cardiovasc Interv. 2010 Feb;3(2):221-9. doi: 10.1016/j.jcin.2009.10.025. PMID 20170881
- [Background] Violi F, Cangemi R. Antioxidant supplements and cardiovascular disease in men. JAMA. 2009 Apr 1;301(13):1335; author reply 1336-7. doi: 10.1001/jama.2009.314. No abstract available. PMID 19336704
- [Background] Cangemi R, Angelico F, Loffredo L, Del Ben M, Pignatelli P, Martini A, Violi F. Oxidative stress-mediated arterial dysfunction in patients with metabolic syndrome: Effect of ascorbic acid. Free Radic Biol Med. 2007 Sep 1;43(5):853-9. doi: 10.1016/j.freeradbiomed.2007.06.002. Epub 2007 Jun 13. PMID 17664149
- [Background] Basili S, Pignatelli P, Tanzilli G, Mangieri E, Carnevale R, Nocella C, Di Santo S, Pastori D, Ferroni P, Violi F. Anoxia-reoxygenation enhances platelet thromboxane A2 production via reactive oxygen species-generated NOX2: effect in patients undergoing elective percutaneous coronary intervention. Arterioscler Thromb Vasc Biol. 2011 Aug;31(8):1766-71. doi: 10.1161/ATVBAHA.111.227959. Epub 2011 Jun 2. PMID 21636808
- [Background] Basili S, Tanzilli G, Raparelli V, Calvieri C, Pignatelli P, Carnevale R, Dominici M, Placanica A, Arrivi A, Farcomeni A, Barilla F, Mangieri E, Violi F. Aspirin reload before elective percutaneous coronary intervention: impact on serum thromboxane b2 and myocardial reperfusion indexes. Circ Cardiovasc Interv. 2014 Aug;7(4):577-84. doi: 10.1161/CIRCINTERVENTIONS.113.001197. Epub 2014 Jul 29. PMID 25074252
- [Result] Pignatelli P, Tanzilli G, Carnevale R, Di Santo S, Loffredo L, Celestini A, Proietti M, Tovaglia P, Mangieri E, Basili S, Violi F. Ascorbic acid infusion blunts CD40L upregulation in patients undergoing coronary stent. Cardiovasc Ther. 2011 Dec;29(6):385-94. doi: 10.1111/j.1755-5922.2010.00168.x. Epub 2010 Jul 12. PMID 20629665